CLINICAL TRIAL: NCT00003615
Title: A Phase II Study of DAB 389 IL-2, an Interleukin-2 Fusion Toxin, for Previously Treated Stage II, III, and IV Follicular Low-Grade Non-Hodgkin's Lymphoma
Brief Title: Denileukin Diftitox in Treating Patients With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Group Chair, Eastern Cooperative Oncology Group
Purpose: Treatment
Other Study IDs: CDR0000066692; E1497
Record Dates: First submitted 1999-11-01; First posted 2004-02-20 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Lymphoma
Keywords: Waldenstrom macroglobulinemia; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse large cell lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse large cell lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse large cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse large cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — denileukin diftitox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: denileukin diftitox

SUMMARY:
RATIONALE: Immunotoxins such as denileukin diftitox can locate cancer cells and kill them without harming normal cells. This may be an effective treatment for non-Hodgkin's lymphoma.

PURPOSE: Phase II trial to study the effectiveness of denileukin diftitox in treating patients who have non-Hodgkin's lymphoma that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response rate in patients with previously treated stage I, II, III, or IV low- or intermediate-grade B-cell non-Hodgkin's lymphoma treated with denileukin diftitox. II. Determine the time to progression, duration of remission, and time to treatment failure in patients after treatment with this therapy. III. Determine the toxicity of this therapy in these patients. IV. Correlate the results of the inteleukin-2 receptor assay with treatment outcomes in these patients.

OUTLINE: Patients are stratified according to interleukin-2 receptor classification (positive vs negative). Patients receive immunotoxin therapy with denileukin diftitox IV over 15-60 minutes on days 1-5. Treatment repeats every 21 days for 2-6 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 33 patients will be accrued for the interleukin-2 (IL-2) receptor-positive stratum and a total of 11-44 patients will be accrued for the IL-2 receptor-negative stratum.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage I, II, III, or IV low- or intermediate-grade B-cell non-Hodgkin's lymphoma Small lymphocytic Follicular small cleaved cell Follicular mixed cell Follicular large cell Marginal Diffuse large B-cell Lymphoplasmacytoid Patients with small lymphocytic lymphoma must have an absolute lymphocyte count less than 10,000/mm3 At least one bidimensionally measurable site At least 1.5 cm in its greatest dimension Not in field of prior radiotherapy Progressive disease after at least one prior treatment regimen for lymphoma A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: See Disease Characteristics Absolute neutrophil count at least 1000/mm3 Platelet count at least 50,000/mm3 Hemoglobin at least 8 g/dL Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) ALT or AST no greater than 2 times ULN Albumin greater than 3.0 g/dL No hepatitis B or C infection Renal: Creatinine no greater than ULN Other: Not pregnant or nursing Fertile patients must use effective contraception HIV negative No active infection requiring anti-infective therapy No other prior invasive malignancy within past 5 years, except: Curatively treated basal cell or squamous cell skin cancer Carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior stem cell transplantation allowed At least 4 weeks since prior biologic therapy No other concurrent immunotherapy Chemotherapy: At least 4 weeks since prior chemotherapy No concurrent chemotherapy Endocrine therapy: At least 4 weeks since prior endocrine therapy No concurrent hormonal therapy (except contraceptives and replacement steroids) No concurrent corticosteroids Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy for localized disease No concurrent radiotherapy Surgery: Not specified Other: No other concurrent experimental medications (including approved drugs tested in an investigational setting)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 1999-05-20 (Actual); Primary Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M. Kuzel, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (10):
- United States (10):
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Trinitas Hospital - Jersey Street Campus, Elizabeth, New Jersey
  - Hunterdon Regional Cancer Center, Flemington, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Riverview Medical Center - Booker Cancer Center, Red Bank, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania

REFERENCES:
- [Result] Kuzel TM, Li S, Eklund J, Foss F, Gascoyne R, Abramson N, Schwerkoske JF, Weller E, Horning SJ. Phase II study of denileukin diftitox for previously treated indolent non-Hodgkin lymphoma: final results of E1497. Leuk Lymphoma. 2007 Dec;48(12):2397-402. doi: 10.1080/10428190701694186. Epub 2007 Oct 13. PMID 17943599